CLINICAL TRIAL: NCT01495884
Title: A Phase I/II Study of Lapatinib Plus Myocet TM in Patients With HER2+ve Metastatic Breast Cancer Following Disease Progression During, or After, Treatment With Trastuzumab and Taxanes
Brief Title: The Myocet/Lapatinib Study. ICORG 10-03, V5
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slower than anticipated accrual
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICORG 10-03
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Her2 Positive Metastatic Breast Cancer
MeSH Terms: interventions — Doxorubicin; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lapatinib (Tyverb™) and (Myocet™) (Experimental)
  Interventions: Drug: non-pegylated liposomal doxorubicon (Myocet™); Drug: Lapatinib (Tyverb™)

INTERVENTIONS:
Drug: non-pegylated liposomal doxorubicon (Myocet™)
Drug: Lapatinib (Tyverb™)

SUMMARY:
This study is a Phase I/II open label, multi-centre trial. Patients with HER2+ve metastatic breast cancer, following disease progression during, or after, treatment with trastuzumab and taxanes, will be treated with Lapatinib (Tyverb™ 500-1250 mg orally daily - depending on the maximum tolerated dose (MTD) determined in the Phase I part of the study) plus Myocet™, 50-60 mg/m2 i.v q3 weeks).

Within the Phase I part, doses are assigned at registration according to the dose escalation scheme.

The dose for the Phase II part of the trial will be based on the MTD established in the Phase I part of the study.

Clinical and laboratory parameters will be assessed to evaluate disease response and toxicity of study therapy. Safety assessments will be performed every 3 weeks for the first 24 weeks. Efficacy assessments (radiological examination) will be performed on all patients every 8 weeks (± 7 days) for the first 24 weeks. Cardiotoxicity assessments will be performed at weeks 6 and 12. From week 24, safety, efficacy and cardiotoxicity assessments will be performed every 12 weeks and at the end of treatment (disease progression, unacceptable toxicity or patient withdraws consent).

DETAILED DESCRIPTION:
Primary Objective:

1. To determine the optimal dose for lapatinib plus Myocet™, in combination, in patients with HER2-positive metastatic breast cancer following disease progression during, or after, treatment with trastuzumab and taxanes (Phase I).
2. To evaluate the 6 month progression-free survival of patients with HER2-positive metastatic breast cancer, following disease progression during, or after, treatment with trastuzumab and taxanes, who are treated with lapatinib plus Myocet™ (Phase II plus patients treated at MTD in Phase I).

Secondary Objectives:

1. To evaluate the overall survival time, duration of progression -free survival, time to treatment failure, confirmed tumour response rate and duration of response in patients treated with this regimen (Phase II plus patients treated at MTD in Phase I).
2. To assess the safety and tolerability of this regimen in these patients.
3. To assess the incidence of cardiotoxicity in these patients treated with this regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedures.
2. Female patients, age ≥ 18 years, who are either post menopausal (post-menopausal status will be defined as patients who are amenorrheic for > 1 year or for a shorter duration if FSH, LH and/or oestradiol levels are within the post-menopausal range), surgically sterile or practicing an effective method of birth control agreed with the patients study physician. Women of childbearing potential should use an effective contraceptive ( such as non hormonal intra uterine device (IUD), condoms, sexual abstinence or vasectomised partner).during treatment and up to 6 months following discontinuation of therapy.
3. Histologically confirmed metastatic breast cancer
4. Documented HER2 overexpression (IHC 3+ or FISH or CISH positive)
5. At least one measurable lesion according to RECIST criteria. Patients with bone only disease are not eligible.
6. Patients with controlled brain metastasis are eligible.
7. Documented disease progression. Progression for entry is defined as appearance of any new lesion not previously identified or increase of 25% or more in existent lesion from previous CT scan and must be documented
8. Prior treatment must have contained trastuzumab and taxane. Patients may have been treated with Lapatinib previously.
9. Life expectancy of at least 12 weeks
10. ECOG Performance Status of ≤ 2
11. Left ventricular ejection fraction (LVEF) ≥ 55%, as measured by Echocardiogram or MUGA Scan (within 14 days prior to first infusion), and no documented history of uncontrolled or symptomatic angina, arrhythmias or congestive heart failure within the previous 6 months
12. Adequate bone marrow, haematological, hepatic and renal function defined as:

    * Absolute Neutrophils Count ≥ 1.5 x 109/L
    * Platelet Count ≥ 100 x 109/L
    * Haemoglobin ≥ 9.0 g/dL
    * Calculated creatinine clearance ≥ 40 mL/min
    * Total bilirubin ≤ ULN. Patients with Gilbert's syndrome prior to study entry must have total bilirubin < 3 x ULN.
    * Alkaline Phosphatase and AST or ALT within the parameters specified in protocol
13. Patients must have recovered from clinically significant side effects associated with prior radiotherapy and chemotherapy
14. Able to swallow and retain oral medication.
15. Formalin-fixed paraffin-embedded tissue from archived tumour tissue samples available (from the primary or metastatic tissue.

Patients meeting any of the following exclusion criteria are not eligible for enrolment into this study:

Exclusion Criteria:

1. Pregnant or lactating women
2. Prior anthracycline chemotherapy with a lifetime dose exceeding 360 mg/m2 doxorubicin or 550 mg/m2 epirubicin
3. Documented history of poorly controlled hypertension), arrhythmia, clinically significant valvular disease, angina requiring treatment, transmural infarction, myocardial infarction within the previous 6 months
4. Concurrent disease that would make the patient inappropriate for study participation, or any other serious medical disorder that would interfere with the patient's safety
5. Dementia, altered mental status, or any other psychiatric condition that would interfere with the patient's safety or informed consent
6. Active or uncontrolled bacterial, viral or fungal infection.
7. History of other malignancy. However patients who have been disease free for 5 years, or patients with a history of resected non-melanoma skin cancer or successfully treated in situ cancer are eligible
8. Concurrent cancer therapy (chemotherapy, immunotherapy, biologic therapy, hormonal therapy, or within 4 weeks preceding the first dose of investigational product)
9. Unresolved or unstable, serious toxicity from prior administration of another investigational product
10. Concurrent treatment with an investigational drug within 4 weeks preceding the first dose of investigational product
11. Known hypersensitivity to lapatinib and Myocet™ or their excipients
12. Any other contraindications for lapatinib and Myocet™
13. Receive concurrent treatment with prohibited medications. Zometa for patients with bone metastasis is allowed. If the patient is on Zometa at start of the study, it should be continued throughout the duration of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Optimal dose for lapatinib plus myocet | 6 months
  Determination of the optimal dose for lapatinib plus Myocet™, in combination, in patients with HER2-positive metastatic breast cancer following disease progression during, or after, treatment with trastuzumab and taxanes as measured by MTD (Phase I)

SECONDARY OUTCOMES:
Overall survival | From registration to death
  overall survival time (OS - time from registration to death from any cause) as assessed by standard RECIST criteria

CONTACTS AND LOCATIONS:
Locations (10):
- Ireland (10):
  - Bon Secours Hospital, Cork
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Mater Misercordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St James's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Limerick, Limerick
  - Waterford Regional Hospital, Waterford